CLINICAL TRIAL: NCT07164092
Title: Efficacy of Topical Atropine Eye Drops for Control of Myopia Progression Among Children Attending Mansoura University Ophthalmic Center
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ghada Allam, Lecturer of Ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Atropine ED for Myopia in MOC
Record Dates: First submitted 2025-08-22; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Atropine, Myopia, Axial elongation
MeSH Terms: conditions — Myopia | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Each participant will receive one drop of atropine 0.05% in one randomly assigned eye and one drop of placebo in the fellow eye nightly for 24 months. No other myopia control treatments will be permitted during the study period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study medications (atropine 0.05% and placebo) will be supplied in identical bottles with identical labeling and packaging to maintain blinding. The allocation of treatment to the right or left eye will be randomized and concealed. Participants, their parents/guardians, the treating investigators, and outcome assessors will remain blinded to the allocation throughout the study. Only the study pharmacist (not involved in outcome assessment) will have access to the randomization code until study completion or unless unmasking is required for safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atropine 0.05% Eye (Experimental): The randomized eye will receive one drop of atropine sulphate 0.05% nightly for 24 months.
  Interventions: Drug: Atropine 0.05% Eye drops
- Placebo Eye (Placebo Comparator): The fellow eye will receive one drop of placebo (vehicle solution without active drug) nightly for 24 months.
  Interventions: Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: Atropine 0.05% Eye drops — The randomized eye will receive one drop of atropine sulphate 0.05% nightly for 24 months.
  Arms: Atropine 0.05% Eye
Drug: Placebo ophthalmic solution — The fellow eye will receive one drop of placebo (vehicle solution without active drug) nightly for 24 months.
  Arms: Placebo Eye

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy and safety of low-dose topical atropine sulphate (0.05%), a non-selective muscarinic antagonist, in slowing the progression of myopia and ocular axial elongation in children. The study will be conducted at Mansoura Ophthalmic Center, Mansoura University, Egypt, from October 2025 to october 2027.

Eligible participants are myopic children attending the outpatient clinic during the study period. Participants will be stratified into three groups according to baseline myopia severity (low, moderate, and high). Each child will be randomized to receive one drop of atropine 0.05% in one eye and one drop of placebo in the fellow eye nightly for 24 months. The allocation of treatment to right or left eye will be randomized to avoid laterality bias.

Study Outcomes

* Primary Outcome

  o Change in ocular axial length (AL) from baseline to 24 months, measured with a NIDEK AL-scan optical biometer (average of five readings within a deviation of ≤0.05 mm). This parameter was used for sample size estimation.
* Secondary Outcomes

  * Change in spherical equivalent refraction (SER), measured by cycloplegic autorefraction using a Topcon KR-800 autorefractor after standard cycloplegia with cyclopentolate 1%.
  * Best-corrected distance visual acuity (BCVA).
* Sample Size

The primary endpoint of this trial is the change in ocular axial length (AL) over 24 months, analyzed as a paired comparison between the atropine-treated and placebo-treated eyes within each child.

Sample size estimation was based on previously published data reporting mean axial elongation of 0.115 ± 0.11 mm in atropine-treated eyes compared with 0.303 ± 0.12 mm in placebo-treated eyes, yielding a mean difference of 0.188 mm. Assuming an inter-eye correlation of 0.6, the standard deviation of the paired difference is estimated at approximately 0.10 mm, giving an effect size of d = 1.88. Using a two-tailed paired t-test with α = 0.05 and 90% power, the minimum required sample size is 12 children.

ELIGIBILITY:
Inclusion Criteria:

* Myopia of at least -1.0 D in both eyes, astigmatism of less than 2.0 D, anisometropia of objective spherical equivalent ≤ 1.50 D.
* Documented myopic progression of at least 0.5 D in the past one year.

Exclusion Criteria:

* Children with ocular or systemic diseases that potentially influence myopia or refractive power.
* Ocular diseases, e.g., cataracts, glaucoma
* Posterior segment hereditary and acquired pathological disorders.
* History of any previous ocular surgery.
* History of any ocular injuries.
* Previous use of interventions (such as atropine, pirenzepine, orthokeratology lens, or other optical methods) for myopia control
* Allergy to atropine, cyclopentolate or benzalkonium chloride

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in ocular axial length (AL) | 2 years
  Change in ocular axial length (AL) from baseline to 24 months, measured with a NIDEK AL-scan optical biometer (average of five readings within a deviation of ≤0.05 mm). This parameter was used for sample size estimation

SECONDARY OUTCOMES:
Change in spherical equivalent refraction (SER | 24 months
  Change in spherical equivalent refraction (SER), measured by cycloplegic autorefraction using a Topcon KR-800 autorefractor after standard cycloplegia with cyclopentolate 1%.
Best-corrected distance visual acuity (BCVA). | 24 months

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided yet